CLINICAL TRIAL: NCT00629798
Title: A Phase II Trial of Busulfan, Melphalan, and Fludarabine With Peri-transplant Palifermin, Followed by a T-Cell Depleted Hematopoietic Stem Cell Transplant From HLA Matched or Mismatched Related or Unrelated Donors in Patients With Advanced Myelodysplastic Syndromes (MDS) and Acute Myeloid Leukemia (AML)
Brief Title: Busulfan, Melphalan, and Fludarabine With Peri-transplant Palifermin, Followed by a T-Cell Depleted Hematopoietic Stem Cell Transplant From HLA Matched or Mismatched Related or Unrelated Donors in Patients With Advanced Myelodysplastic Syndromes (MDS) and Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-008
Record Dates: First submitted 2008-02-14; First posted 2008-03-06 (Estimated); Results first posted 2021-09-24 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2020-10

CONDITIONS: Acute Myeloid Leukemia; Advanced Myelodysplastic Syndromes
Keywords: Busulfan; Melphalan; Fludarabine; 08-008
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Busulfan; Melphalan; fludarabine; Antilymphocyte Serum; Fibroblast Growth Factor 7; Stem Cell Transplantation; Guidelines as Topic

ARMS (1):
- 1 (Experimental): This is a single arm phase II trial to assess the efficacy (decrease the transplant related mortality) and safety of peri-transplant Palifermin in combination with a preparative regimen with busulfan, melphalan, fludarabine, and anti-thymocyte globulin (ATG), and a T cell depleted stem cell transplant from a histocompatible related or unrelated donor in patients with advanced MDS and AML evolved from MDS. The addition of Palifermin is to decrease the toxicity and the infection rate associated with this regimen and transplant type and to foster earlier immune reconstitution.
  Interventions: Drug: Busulfan, Melphalan, Fludarabine, Anti-Thymocyte Globulin, Palifermin, Stem cell transplant

INTERVENTIONS:
Drug: Busulfan, Melphalan, Fludarabine, Anti-Thymocyte Globulin, Palifermin, Stem cell transplant — Patients will receive Palifermin 60 mcg/kg/day IV on three consecutive days with the last dose administered no less than 24 and no more than 48 hr prior to start of cytoreduction. The preparative regimen to be used for transplants will consist: of busulfan administered in 12 doses over three days of 0.8 mg/kg IV for patients > or = to 4 years of age or 1.0 mg/kg IV for patients < 4 years of age; melphalan 70 mg/m2 IV x 2 days; and, fludarabine 25 mg/m2 IV x 5 days
  Other Names: Patients will receive ATG for two doses prior to transplant.; G-CSF mobilized CD34+E- PBSCs (or BM if donors are unwilling or unable; to donate PBSC) obtained from the HLA compatible donor will be infused on; day 0. Patients will receive three additional daily doses of Palifermin,; the first approximately 6 hours after the stem cell infusion on day 0,; followed by two daily doses given on d+1 and d+2. Supportive care will be administered as per the BMT Service; guidelines.

SUMMARY:
This study will see if the researchers can lower that risk by giving the patient Palifermin. This drug helps protect the lining of the mouth, throat, and stomach. These areas typically get sores or ulcers while the blood cell counts are very low. The patient can get infections in or from these sores. Palifermin might also help the immune system recover faster. It is currently approved for patients who receive their own stem cells. That is called an autologous transplant. This study will test the use of Palifermin for T-cell depleted allogeneic stem cell transplants.

ELIGIBILITY:
Inclusion Criteria:

* Patients should be < 65 years. Patients > or equal to 65 years will be accrued on a case by case basis after discussion and approval by the BMT Service.
* Patients may be of either gender or any ethnic background.
* Patients must have a Karnofsky or Lansky Performance Status > or equal to 70%.
* Patients must have adequate organ function measured by:

  * Cardiac: asymptomatic or if symptomatic then LVEF at rest must be > or equal to 50% and must improve with exercise.
* Hepatic: < 3x ULN ALT and < 1.5 total serum bilirubin, unless there is congenital benign hyperbilirubinemia.

  * Renal: serum creatinine < than or equal to 1.2 mg/dl or if serum creatinine is outside the normal range, then CrCl > 60-ml/min/1.73 m2
  * Pulmonary: asymptomatic or if symptomatic, DLCO > 50% of predicted (corrected for hemoglobin)
* Each patient must be willing to participate as a research subject and must sign an informed consent form.
* Parent or legal guardians of patients who are minors will sign the informed consent form.

Exclusion Criteria:

* Active CNS or skin leukemic involvement
* Female patients who are pregnant or breast-feeding
* Active viral, bacterial or fungal infection
* Patient seropositive for HIV-I/II; HTLV -I/II
* Patients who have undergone a prior allogeneic or autologous stem cell transplant within the previous six months.
* Patients who have had a previous malignancy that is not in remission.

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2008-02-12 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2020-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roni Tamari, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Palifermin: This is a single arm phase II trial to assess the efficacy (decrease the transplant related mortality) and safety of peri-transplant Palifermin in combination with a preparative regimen with busulfan, melphalan, fludarabine, and anti-thymocyte globulin (ATG), and a T cell depleted stem cell transplant from a histocompatible related or unrelated donor in patients with advanced MDS and AML evolved from MDS. The addition of Palifermin is to decrease the toxicity and the infection rate associated with this regimen and transplant type and to foster earlier immune reconstitution.
  Busulfan, Melphalan, Fludarabine, Anti-Thymocyte Globulin, Palifermin, Stem cell transplant: Patients will receive Palifermin 60 mcg/kg/day IV on three consecutive days with the last dose administered no less than 24 and no more than 48 hr prior to start of cytoreduction. The preparative regimen to be used for transplants will consist: of busulfan administered in 12 doses over three days of 0.8 mg/kg IV for patients > or = to 4 years of age or 1.0 mg/kg IV for patients < 4 years of age; melphalan 70 mg/m2 IV x 2 days; and, fludarabine 25 mg/m2 IV x 5 days
Period: Overall Study
Arm/Group | Palifermin
Started | 64
Completed | 60
Not Completed | 4
Not completed — Not Treated | 4

BASELINE CHARACTERISTICS:
Arm/Group | Palifermin
Number analyzed (Participants) | 64
Age, Continuous [Median (Full Range); unit: years] | 60 [4 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 61
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 58
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 64

OUTCOME MEASURES:

1. Primary Outcome: To Reduce the Early Transplant-related Mortality.
Time Frame: conclusion of study
Population: Data were not collected
Arm/Group | Palifermin
Number analyzed (Participants) | 0

2. Secondary Outcome: To Improve the Quality of Immune Reconstitution Following Transplantation.
Time Frame: conclusion of study
Population: Data were not collected
Arm/Group | Palifermin
Number analyzed (Participants) | 0

3. Secondary Outcome: To Reduce the Incidence Rate of Fatal Post Transplant Infectious Complications.
Time Frame: conclusion of study
Population: Data were not collected
Arm/Group | Palifermin
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Palifermin
All-Cause Mortality (participants affected / at risk) | 38/64
Serious Adverse Events (participants affected / at risk) | 28/64
Other Adverse Events (participants affected / at risk) | 28/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Palifermin (N=64)
Acidosis (metabolic/respiratory) (Metabolism and nutrition disorders) | 1
Adult Respiratory Distress Synd (ARDS) (Respiratory, thoracic and mediastinal disorders) | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 1
Bilirubin (hyperbilirubinemia) (Investigations) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Death not assoc w CTCAE term - Death NOS (General disorders) | 4
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Fever (in the absence of neutropenia) (General disorders) | 1
Hemorrhage, Upper GI NOS (Gastrointestinal disorders) | 1
Hemorrhage/Bleeding, other (Blood and lymphatic system disorders) | 1
Hypotension (Vascular disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 11
Inf norm ANC/gr1/2 neut-Pneumonia (lung) (Infections and infestations) | 3
Infection, other (Infections and infestations) | 10
Liver dysfunction/failure (Renal and urinary disorders) | 2
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 2
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 1
Pain - Sinus (Respiratory, thoracic and mediastinal disorders) | 1
Platelets (Investigations) | 1
Pleural effusion (non-malig) (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis/pulm inflitrates (Respiratory, thoracic and mediastinal disorders) | 1
Pulm/upp respiratory - Other (spec) (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2
Renal failure (Renal and urinary disorders) | 1
Renal/Genitourinary-Other Specify (Renal and urinary disorders) | 3
Seizure (Nervous system disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Palifermin (N=64)
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 26
ALT, SGPT (Investigations) | 21
Creatinine (Investigations) | 18
Magnesium, high (hypermagnesemia) (Metabolism and nutrition disorders) | 14
AST/SGOT (Investigations) | 12
Bilirubin (hyperbilirubinemia) (Investigations) | 10
Alkaline phosphatase (Investigations) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-02): https://cdn.clinicaltrials.gov/large-docs/98/NCT00629798/Prot_SAP_000.pdf